CLINICAL TRIAL: NCT04271150
Title: Clinical Evaluation of Universal Adhesive's Different Application Modes
Brief Title: Efficiency of Different Modes of Universal Adhesive
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Zeynep Bilge Kutuk, Assistant Professor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KA-180016
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Dental Caries; Adhesion
MeSH Terms: conditions — Dental Caries; Tissue Adhesions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-etch (Experimental): Self-etch mode of the universal adhesive will be used
  Interventions: Device: Self-etch
- Total-etch (Active Comparator): Total etch mode of the universal adhesive will be used
  Interventions: Device: Total-etch

INTERVENTIONS:
Device: Self-etch — Universal adhesive with self-etch mode
  Arms: Self-etch
Device: Total-etch — Universal adhesive with total-etch mode
  Arms: Total-etch

SUMMARY:
The purpose of this study is to evaluate and compare the clinical performance of a Universal adhesive's different application modes.

DETAILED DESCRIPTION:
Class 2 composite restorations will be placed using a bulk-fill composite resin restorative on two posterior teeth with proximal caries, in a split mouth design. 25 patients will be included in the study. The teeth will be randomized into two groups according to the application mode of universal adhesive material.

Group 1: the universal adhesive will be used in etch-and-rinse mode Group 2: the universal adhesive will be used in self-etch mode. The US Public Health Service criteria (secondary caries, anatomical form, surface roughness, marginal integrity, marginal discoloration and retention) will be used for clinical evaluation of atraumatic resin restorations. The restorations will be evaluated at baseline and 6th, 12th, 18th, 24th months. Intra-oral photos will be taken directly after treatment and at control appointments to evaluate discoloration and seconder caries under magnification.

The data will be analysed statistically using Fisher's Exact Test; and the Kaplan-Meier and Wilcoxon method will be used to estimate survival percentages.

ELIGIBILITY:
Inclusion Criteria:

* a need for at least two but not more than four posterior tooth-colored restorations
* the presence of teeth to be restored in occlusion
* teeth that were symptomless and vital
* a normal periodontal status
* a good likelihood of recall availability.

Exclusion Criteria:

* partly erupted teeth
* absence of adjacent and antagonist teeth
* poor periodontal status
* adverse medical history
* potential behavioral problems

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Marginal adaptation | From baseline to 6 year the change of restorations will be evaluated
  Observers will evaluate the restorations will be performed using the modified United State Public Health Service criteria regarding marginal adaptation.
  Marginal adaptation will evaluated by 2 independent clinicians. Visual inspection with a mirror at 18 inches will be performed . A score means the higher score of clinical acceptability while C and D score means that the restoration has failed and needs to be replaced. Alpha 1: Harmonious outline Alpha 2: Marginal gap (max 100μ) with discoloration (removable) Bravo: Marginal gap (> 100μ) with discoloration (unremovable) Charlie: The restoration is fractured or missed.
Marginal discoloration | From baseline to 6 year the change of restorations will be evaluated
  Observers will evaluate the restorations will be performed using the modified United State Public Health Service criteria regarding marginal discoloration.
  Marginal discoloration will be evaluated by 2 independent clinicians. Visual inspection with a mirror at 18 inches will be performed . A score means the higher score of clinical acceptability while C score means that the restoration has failed and needs to be replaced. Alpha: No discoloration anywhere along the margin between the restoration and the adjacent tooth. Bravo: Slight discoloration along the margin between the restoration and the adjacent tooth. Charlie: The discoloration penetrated along the margin of the restorative material in a pulpal direction.
Retention | From baseline to 6 year the change of restorations will be evaluated.
  Observers will evaluate the restorations will be performed using the modified United State Public Health Service criteria regarding retention rate.
  Retention rate will be evaluated by 2 independent clinicians. Visual inspection with a mirror at 18 inches was performed . A score means the higher score of clinical acceptability while C and D score means that the restoration has failed and needs to be replaced. Alpha 1:Clinically excellent Alpha 2: Clinically good with slight deviations from ideal performance, correction possible without damage of tooth or restoration Bravo: Clinically sufficient with few defects, corrections or repair of the restoration possible Charlie: Restoration is partially missed Delta: Restoration is totally missed
Anatomic form | From baseline to 6 year the change of restorations will be evaluated.
  Observers will evaluate the restorations will be performed using the modified United State Public Health Service criteria regarding anatomic form.
  Anatomic form will be evaluated by 2 independent clinicians. Visual inspection with a mirror at 18 inches was performed . A score means the higher score of clinical acceptability while C score means that the restoration has failed and needs to be replaced. Alpha 1: Continuous with existing anatomical form Alpha 2: Slightly discontinuous due to some chipping on the proximal ridge Bravo: Discontinuous with existing anatomical form due to material loss but proximal contact still present Charlie: Proximal contact is lost with ridge fracture.
Color change | From baseline to 6 year the change of restorations will be evaluated.
  Observers will evaluate the restorations will be performed using the modified United State Public Health Service criteria regarding color change. Color changes will be evaluated by 2 independent clinicians. Visual inspection with a mirror at 18 inches was performed . A score means the higher score of clinical acceptability while C score means that the restoration has failedand needs to be replaced. Alpha: The restoration matches the adjacent tooth structure in color and translucency. Bravo: Light mismatch in color, shade or translucency between the restoration and the adjacent tooth. Charlie: The mismatch in color and translucency is outside the acceptable range of tooth color and translucency.

CONTACTS AND LOCATIONS:
Overall Officials: Ayse R Yazici, DDS, PhD, Study Director — Hacettepe University School of Dentistry
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: PUBMED — https://www.ncbi.nlm.nih.gov/pubmed/28581919
- See also: PUBMED — https://www.ncbi.nlm.nih.gov/pubmed/29630489